CLINICAL TRIAL: NCT02699281
Title: N-of-1 Randomised Trials to Assess the Efficacy of Ultra-micronized Palmitoylethanolamide (Um-PEA) in Geriatric Patients With Chronic Pain
Brief Title: Efficacy of Ultra-micronized Palmitoylethanolamide (Um-PEA) in Geriatric Patients With Chronic Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Maura Marcucci, MD, MSc, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Nof1-PEA
Record Dates: First submitted 2016-02-21; First posted 2016-03-04 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultra-micronized Palmitoylethanolamide (Experimental): Ultra-micronized Palmitoylethanolamide 600 mg twice a day
  Interventions: Drug: ultra-micronized palmitoylethanolamide
- Placebo (Placebo Comparator): Placebo tab twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ultra-micronized palmitoylethanolamide — ultra-micronized palmitoylethanolamide 600 mg twice a day
  Other Names: um-PEA; Normast
  Arms: Ultra-micronized Palmitoylethanolamide
Drug: Placebo — um-PEA like placebo twice a day
  Other Names: um-PEA like placebo
  Arms: Placebo

SUMMARY:
Investigators planned to adopt the N-of-1 trial approach to objectively test the effectiveness of ultra-micronized PEA at an individual level in our older outpatients. 65 years old or older persons referring to the Geriatric Unit of the Fondazione IRCSS Ca' Granda Ospedale Maggiore Policlinico of Milan complaining of noncancer chronic pain of any origin will be eligible. Each trial will be a placebo-controlled randomized crossover trial including two um-PEA (600 mg twice a day) and placebo treatment pairs. Investigators will secondarily meta-analyse the performed N-of-1 trials to obtain an estimate of the average effect of um-PEA compared with placebo using a frequentist and Bayesian approach.

DETAILED DESCRIPTION:
Background: Chronic pain in the elderly is highly prevalent, often underestimated, and associated with adverse outcomes. Most available analgesic drugs are often either ineffective or not tolerated, and burdened with many side effects. Palmitoylethanolamide (PEA) is an endogenous widely distributed N-acylethanolamina involved in neuroinflammation and pain generating processes. Formulations containing ultra-micronized Palmitoylethanolamide (um-PEA) are available on the market but their effectiveness on chronic pain in highly heterogeneous geriatric patients is not clear and likely not generalizable. Investigators planned to adopt the N-of-1 trial approach to objectively test the effectiveness of ultra-micronized PEA at an individual level in our older outpatients.

Methods/Design: 65 years old or older persons referring to the Geriatric Unit of the Fondazione IRCSS Ca' Granda Ospedale Maggiore Policlinico of Milan complaining of noncancer chronic pain of any origin will be eligible. Each trial will be a placebo-controlled randomized crossover trial including two um-PEA (600 mg twice a day) and placebo treatment pairs. um-PEA or placebo 3-week periods will be separated by 2-week washout intervals to overcome the possible carryover effect. Pain intensity, need for on-demand analgesic medications, and impact on daily activities will be evaluated. Also, cognitively impaired patients will be eligible as long as the expression of pain can be recognized and its frequency assessed by a caregiver. Trial results will be then discussed with the patient/caregiver and the treating physician to decide whether to continue the treatment. The impact of the N-of-1 approach on the physician's management plan and confidence will be assessed. Investigators will secondarily meta-analyse the performed N-of-1 trials to obtain an estimate of the average effect of um-PEA compared with placebo using a frequentist and Bayesian approach.

Discussion: While pursuing an ultimate clinical objective, i.e. to empirically and objectively decide the best treatment choice for an individual older patient with chronic pain, these series of geriatric N-of-1 trials on PEA will bring the Evidence Based Medicine principles into the care of patients not usually represented in conventional randomized controlled trials, and realize a patient-centered outcome approach necessary to improve appropriate prescribing in elderly patients with multimorbidity and polypharmacy.

ELIGIBILITY:
Inclusion Criteria:

* Pain is located at the back (any level) and/or at the joints and/or at the limbs.
* The pain is chronic, i.e. it has been present for at least 6 months, even if with fluctuations.
* The pain is attributable to one or more of the following conditions: osteoarthritis/osteoarthrosis; spondylosis; radiculopathy; diabetic peripheral neuropathy; post-herpetic neuralgia; chronic idiopathic axonal polyneuropathy; fibromyalgia; or pain of uncertain origin or idiopathic, as long as it has had and it is expected to have a chronic nature, even if with spontaneous fluctuations.

Exclusion Criteria:

* cancer-related pain
* clear ischemic pathogenesis for pain (e.g. claudicatio intermittens or critical limb ischemia)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
daily intensity of pain assessed using a 11-point visual numeric scale, accompanied with labels and pictures, modified from Faces Pain Scale. | 126 days

SECONDARY OUTCOMES:
daily need of on-demand analgesic medications | 126 days
impact of pain on daily activities (short questionnaire modified from the back pain functional scale) | 126 days
  The short questionnaire modified from the back pain functional scale consists of 12 items (but it can be modified to better fit to the patients). A score from 1 to 5 is assigned to each item.

CONTACTS AND LOCATIONS:
Overall Officials: Maura Marcucci, MD, MSc, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Geriatric Unit, Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Germini F, Coerezza A, Andreinetti L, Nobili A, Rossi PD, Mari D, Guyatt G, Marcucci M. N-of-1 Randomized Trials of Ultra-Micronized Palmitoylethanolamide in Older Patients with Chronic Pain. Drugs Aging. 2017 Dec;34(12):941-952. doi: 10.1007/s40266-017-0506-2. PMID 29210011
- [Derived] Marcucci M, Germini F, Coerezza A, Andreinetti L, Bellintani L, Nobili A, Rossi PD, Mari D. Efficacy of ultra-micronized palmitoylethanolamide (um-PEA) in geriatric patients with chronic pain: study protocol for a series of N-of-1 randomized trials. Trials. 2016 Jul 29;17:369. doi: 10.1186/s13063-016-1496-9. PMID 27473188